CLINICAL TRIAL: NCT03640923
Title: Study of the Germinal Transmission After Endogenization of HIV Sequences Without a Competent Virus for Replication and a Potential Protective Role
Brief Title: Germinal Transmission After Endogenization of HIV Sequences Without a Competent Virus for Replication and a Potential Protective Role
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-23
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Child with a proven infection of the mother or both biological parents known to HIV antenatal a swab of mucous membrane will be withdrawed
  Interventions: Other: a swab of mucous membrane

INTERVENTIONS:
Other: a swab of mucous membrane — a swab of mucous membrane in oredre to analyse the genome

SUMMARY:
It is necessary to better understand the transmission of human immunodeficiency virus (HIV) genome sequences by gametes without replication-competent virus transmission. In fact, HIV endogenization could be protective. Some studies are supporting this hypothesis, one shew the presence of HIV genome sequences in spermatozoa, and others show that HIV-positive "Elite controllers" patients have HIV genome sequences without a replication competent virus. One study found HIV genome sequences without a replication-competent virus in the cells of an HIV-negative child whose mother is a non-sick HIV-positive. We will conduct a prospective descriptive and analytical study over a period of 2 years, from September 2018 to November 2020. We will explore by FISH method in the IHU Méditerranée-Infection laboratory, Marseille, the presence or absence of HIV genome sequences without a replication-competent virus in epithelial cells of children with parents are infected by HIV. Children included must be under 12 months of age, followed at Robert Debré Hospital, Paris or Timone Enfant Hospital, Marseille because of a parental HIV infection. They must have the recommended blood tests to assess their HIV status and the parents consent should be written. Subsequent progression to HIV infection or not will be followed and a statistical study will be conducted to establish a link between the presence of endogenized HIV genome sequences in epithelial cells and the developpement or not of HIV infection.

DETAILED DESCRIPTION:
It is necessary to better understand the transmission of human immunodeficiency virus (HIV) genome sequences by gametes without replication-competent virus transmission. In fact, HIV endogenization could be protective. Some studies are supporting this hypothesis, one shew the presence of HIV genome sequences in spermatozoa, and others show that HIV-positive "Elite controllers" patients have HIV genome sequences without a replication competent virus. One study found HIV genome sequences without a replication-competent virus in the cells of an HIV-negative child whose mother is a non-sick HIV-positive. We will conduct a prospective descriptive and analytical study over a period of 2 years, from September 2018 to November 2020. We will explore by FISH method in the IHU Méditerranée-Infection laboratory, Marseille, the presence or absence of HIV genome sequences without a replication-competent virus in epithelial cells (non-hematogenous) of children with parents are infected by HIV. Children included must be under 12 months of age, followed at Robert Debré Hospital, Paris or Timone Enfant Hospital, Marseille because of a parental HIV infection. They must have the recommended blood tests to assess their HIV status and the parents consent should be written. Subsequent progression to HIV infection or not will be followed and a statistical study will be conducted to establish a link between the presence of endogenized HIV genome sequences in epithelial cells and the developpement or not of HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Children included must be under 12 months of age

  * Followed at Robert Debré Hospital, Paris or Timone Enfant Hospital, Marseille
  * Parental HIV infection
  * They must have the recommended blood tests to assess their HIV status
  * Parents consent should be written

Exclusion Criteria:

* Absence of parents consents

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Number of child with HIV genome sequences | 1 day
  Presence or absence of HIV genome sequences within the child's epithelial cells.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France